CLINICAL TRIAL: NCT05188196
Title: Efficacy of Collagen Sponge Versus Collagen Membrane in Combination With Collagenated Bovine Bone Mineral on Ridge Preservation of Compromised Extraction Sockets in Periodontitis Patients: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Collagen Sponge Versus Collagen Membrane on Ridge Preservation of Periodontally Compromised Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Peihui Ding, Principal Investigator, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZhejiangU-2021（77）
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Membrane (Active Comparator): ridge preservation with collagen membrane + collagenated bovine bone mineral
  Interventions: Procedure: alveolar ridge preservation
- Collagen Sponge (Experimental): ridge preservation with collagen sponge + collagenated bovine bone mineral
  Interventions: Procedure: alveolar ridge preservation

INTERVENTIONS:
Procedure: alveolar ridge preservation — Alveolar ridge preservation and augmentation commonly are performed immediately after tooth extraction to preserve or increase ridge volume within or beyond the skeletal envelope that exists at the time of extraction.

SUMMARY:
The study aims to evaluate the efficacy of ridge preservation with collagen sponge or collagen membrane in combination with collagenated bovine bone mineral in extraction sockets of periodontally diseased teeth.

DETAILED DESCRIPTION:
The study aims to evaluate the changes of clinical and radiographic outcomes following ridge preservation with collagen sponge or collagen membrane in combination with collagenated bovine bone mineral in extraction sockets of periodontally diseased teeth. The included patients will be randomized into two groups. The patients in control group will be treated with collagen membrane + collagenated bovine bone mineral, and those in the test group will be treated with collagen sponge + collagenated bovine bone mineral. The horizontal width of ridge, the vertical height of ridge at the buccal and palatal/lingual plates, width of keratinized tissue and thickness of mucosa will be measured before surgery and at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Need for molar extraction due to periodontal disease and plan for late implantation
3. No acute infection, such as abscess or effusion
4. Presence of bone defects on at one or two socket walls, where the height of the horizontal (suprabony) component of the defect (alveolar bone crest - cement-enamel junction) is >50% of the corresponding root length and the bone height of socket walls is at least 3 mm
5. Presence of one adjacent tooth to the extraction site

Exclusion Criteria:

1. Smoking
2. Pregnancy or lactation
3. Untreated periodontal disease
4. Severe systemic conditions that contraindicate surgery (such as diabetes, heart disease, cancer etc.)
5. Under radiotherapy
6. Systemic disease or medication that influences bone metabolism and mucosal healing (such as immunosuppressants, phenytoin, bisphosphonates etc.)
7. Extraction of multiple adjacent teeth
8. Allergy to any of the materials used in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline horizontal width of ridge at 6 months | baseline, at 6 months
  horizontal width of ridge at 1, 3, 5mm below crest
change from baseline vertical height of ridge at 6 months | baseline, at 6 months
  vertical height of ridge at the buccal and palatal/lingual plates

SECONDARY OUTCOMES:
width of keratinized tissue | at 6 months
  measured from the MGJ to the mucosa margin at the mid-buccal aspect using a periodontal probe
thickness of mucosa | at 6 months
  measured at the mid-buccal aspect using an endodontic file with a rubber stop
postoperative pain | at 2 weeks
  using a visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Peihui Ding, Doctor, Principal Investigator — The Affiliated Stomatology Hospital of Zhejiang University School of Medicine
Locations (1):
- The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No